CLINICAL TRIAL: NCT05344872
Title: Automatic Tube Compensation Versus Pressure Support for Ventilatory Weaning of Pediatrics Postcardiac Surgery
Brief Title: ATC Vs PSV for Ventilatory Weaning of Pediatrics Postcardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 193
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-04

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Weaning trial will be done for 17 patients using PSV 0 cmH2O with 100% automatic tube compensation (ATC).
  Interventions: Other: Weaning from mechanical ventilation
- Group B (Active Comparator): Weaning trial will be done for 17 patients using PSV 8 cmH2O without ATC.
  Interventions: Other: Weaning from mechanical ventilation

INTERVENTIONS:
Other: Weaning from mechanical ventilation — Weaning from mechanical ventilation post congenital cardiac surgery

SUMMARY:
The ventilator modality of automatic tube compensation (ATC) can provide variable pressure supports during the weaning process to overcome any change in the resistance of the breathing circuit, endotracheal tube, and airways. The aim of the study is to evaluate the automatic tube compensation (ATC) as a tool for ventilatory weaning in pediatrics after surgeries for congenital cardiac anomalies.

DETAILED DESCRIPTION:
The ventilator modality of automatic tube compensation (ATC) can provide variable pressure supports during the weaning process to overcome any change in the resistance of the breathing circuit, endotracheal tube, and airways. ATC is effective in overcoming the work of breathing caused by airway resistance to allow successful weaning process and extubation. Pressure support ventilation (PSV) has been widely used in the performance of a spontaneous breathing trial because it can compensate to some extent for the additional work of breathing imposed by the endotracheal tube and the breathing circuit. However, it is difficult to recognise the exact pressure support to overcome the tubing resistance during the weaning process till extubation. The aim of the study is to evaluate the automatic tube compensation (ATC) as a tool for ventilatory weaning in pediatrics after surgeries for congenital cardiac anomalies. The primary objective of our study is to compare the efficacy of ATC versus PS as a modality for ventilatory weaning of pediatric postcardiac surgery as regards effects on work of breathing, lung compliance, and alveolar recruitment. The secondary objective is to determine perioperative predictors of extubation failure (requirement for reintubation and mechanical ventilation after prior successful weaning from ventilation, within 48 hours after extubation) after cardiac surgery. Patients will be included after fulfilling weaning criteria and being pain free. a weaning trial for 30 minutes will be commenced according to the following and assessed by the attending physician:- Group A: Weaning trial will be done for 17 patients using PSV 0 cmH2O with 100% automatic tube compensation (ATC).

Group P: Weaning trial will be done for 17 patients using PSV 8 cmH2O without ATC.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients (age 8 months to 12 years) who will undergo congenital cardiac surgeries with the same general anesthetic technique and Pecto-intercostal fascial plane block (PIFB) as regional analgesia for pain management.

Exclusion Criteria:

* (1) Duration of mechanical ventilation is more than 48 hours; (2) Patients on high inotropic support (unstable hemodynamics); (3) Patients with disturbed conscious level; (4) Patients with palliative cardiac shunting procedures (e.g., BT shunt, Glenn shunt).

Ages: 8 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Minute ventilation | 1 year
  Tidal volume (ml/kg) × respiratory rate (breath / minutes)
Oxygenation index (OI) | 1 year
  mean air way pressure × FIO2/PaO2
Work of breathing (WOB) | 1 year
  (∆ V × flow × R + Volume/compliance) (J/L/Kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt